CLINICAL TRIAL: NCT01187238
Title: A Randomized Multicenter Phase II Study of Intensity-modulated Radiotherapy Combined With Chemotherapy Versus Intensity-modulated Radiotherapy Alone for Stage II Nasopharyngeal Carcinoma
Brief Title: The Value of Concurrent Chemoradiotherapy for Stage II Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jun-Lin Yi, MD, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH-HN-001
Record Dates: First submitted 2010-08-18; First posted 2010-08-24 (Estimated); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma; Stage II; Intensity-modulated radiotherapy; Concurrent chemoradiotherapy; Cisplatin
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm1-radical radiotherapy alone group (No Intervention): Arm1-radical radiotherapy alone group, the eligibility patients will received radical intensity-modulated radiotherapy alone
- Arm2-concurrent chemoradiotherapy group (Experimental): Arm2-concurrent chemoradiotherapy group, the eligibility patients will received radiotherapy the same as radical radiotherapy arm,and also will received the concurrent chemotherapy wiht the regimen consist of cisplatin 40mg/m2, weekly for 7weeks.
  Interventions: Drug: cisplatin

INTERVENTIONS:
Drug: cisplatin — in experimental arm, the eligibility patients will be received the same radiotherapy as radical radiotherapy alone group, and also will received concurrent chemotherapy with the regimen of cisplatin 40mg/m2, weekly,from week 1 to week 7
  Other Names: DDP
  Arms: Arm2-concurrent chemoradiotherapy group

SUMMARY:
The purpose of this study is to verify the role of adding cisplatin chemotherapy to the intensity-modulated radiotherapy (IMRT) for stage II nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
Clinical Stage II nasopharyngeal carcinoma consisted of T2N0M0, T1N1M0, T2N1M0 three subgroups, the data came from conventional radiotherapy era showed that the prognosis of this three subgroups were different, the N1 groups suffered more distant metastasis than N0 group, and some literature showed that combined chemotherapy with radiotherapy in stage II patients can improve the treatment results.

Intensity-modulated radiotherapy (IMRT)now is an widely used technique in the treatment of nasopharyngeal carcinoma, the preliminary results showed that IMRT can improve the quality of life in nasopharyngeal through salivary gland preservation.

Compared IMRT alone with IMRT plus cisplatin concurrent chemotherapy in the treatment of stageII nasopharyngeal carcinoma, we hope to confirm whether stage II (and which subgroup) nasopharyngeal carcinoma will be benefit from concurrent chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* pathological confirmed squamous cell carcinoma, WHO II-III type,
* clinical stage II (UICC 7th edition, 2009)
* Karnovsky performance score > 70
* first course of radiotherapy, without radiotherapy and chemotherapy history for other head and neck cancer.
* anticipated life span more than 6 month
* Hemoglobin > 120g/L, WBC > 4.0x10*9/L, Plt > 100x10*9/L
* liver and renal function under the 1.25 normal upper limit
* with written consent information

Exclusion Criteria:

* have other cancer history
* have chemotherapy history
* have radiotherapy history
* have head and neck surgery history(exclusion lymph node biopsy)
* evidence showed distant metastasis or other cancer
* other severe medical comorbidity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2010-05; Primary Completion 2012-07 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Acute toxicities | 2 years
  Acute toxicity will be measured by CTCAE3.0

SECONDARY OUTCOMES:
Long term treatment results | 5 years
  1-, 3-year local-regional control, overall survival, disease-free survival, distant metastasis-free survival will be observed.

CONTACTS AND LOCATIONS:
Overall Officials: Li Gao, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (3):
- China (3):
  - Cancer hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Zhejiang province cancer hospital, Hangzhou, Zhejiang
  - Cancer hospital, Chinese Academy of Medical Sciences, Beijing

REFERENCES:
- [Background] Kam MK, Leung SF, Zee B, Chau RM, Suen JJ, Mo F, Lai M, Ho R, Cheung KY, Yu BK, Chiu SK, Choi PH, Teo PM, Kwan WH, Chan AT. Prospective randomized study of intensity-modulated radiotherapy on salivary gland function in early-stage nasopharyngeal carcinoma patients. J Clin Oncol. 2007 Nov 1;25(31):4873-9. doi: 10.1200/JCO.2007.11.5501. PMID 17971582
- [Background] Chua DT, Sham JS, Kwong DL, Au GK. Treatment outcome after radiotherapy alone for patients with Stage I-II nasopharyngeal carcinoma. Cancer. 2003 Jul 1;98(1):74-80. doi: 10.1002/cncr.11485. PMID 12833458
- [Result] Chua DT, Ma J, Sham JS, Mai HQ, Choy DT, Hong MH, Lu TX, Au GK, Min HQ. Improvement of survival after addition of induction chemotherapy to radiotherapy in patients with early-stage nasopharyngeal carcinoma: Subgroup analysis of two Phase III trials. Int J Radiat Oncol Biol Phys. 2006 Aug 1;65(5):1300-6. doi: 10.1016/j.ijrobp.2006.02.016. Epub 2006 Jun 5. PMID 16750333
- [Result] Cheng SH, Tsai SY, Yen KL, Jian JJ, Chu NM, Chan KY, Tan TD, Cheng JC, Hsieh CY, Huang AT. Concomitant radiotherapy and chemotherapy for early-stage nasopharyngeal carcinoma. J Clin Oncol. 2000 May;18(10):2040-5. doi: 10.1200/JCO.2000.18.10.2040. PMID 10811668
- [Derived] Huang X, Chen X, Zhao C, Wang J, Wang K, Wang L, Miao J, Cao C, Jin T, Zhang Y, Qu Y, Chen X, Liu Q, Zhang S, Zhang J, Luo J, Xiao J, Xu G, Gao L, Yi J. Adding Concurrent Chemotherapy to Intensity-Modulated Radiotherapy Does Not Improve Treatment Outcomes for Stage II Nasopharyngeal Carcinoma: A Phase 2 Multicenter Clinical Trial. Front Oncol. 2020 Aug 7;10:1314. doi: 10.3389/fonc.2020.01314. eCollection 2020. PMID 32850414